CLINICAL TRIAL: NCT00000324
Title: Tryptophan and Behavior Therapy for Cocaine Abuse
Brief Title: Tryptophan and Behavior Therapy for Cocaine Abuse - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Johns Hopkins University (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-10754-1; R01-10754-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2005-08

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Tryptophan

INTERVENTIONS:
Drug: Tryptophan

SUMMARY:
The purpose of this study is to assess the efficacy of tryptophan vs. placebo, and voucher payments vs. a control condition, in the treatment of cocaine dependence.

DETAILED DESCRIPTION:
This clinical trial uses a 2 by 2 design to compare tryptophan to placebo, and voucher incentives vs. a control condition, in the outpatient treatment of cocaine dependence- using a relapse prevention model of treatment intervention.

ELIGIBILITY:
Inclusion Criteria:

* Cocaine dependent

Exclusion Criteria:

* Physically dependent on drugs of abuse other than cocaine
* Significant medical or psychiatric illness (besides substance abuse disorder)
* Pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 1997-03; Study Completion 2001-04

PRIMARY OUTCOMES:
Side effects
Retention
Cocaine use
Cocaine craving
Other drug use
Psychosocial functioning

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Strain, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Jones H.E., Johnson, R.E., Bigelow G.E., Strain E.C. Differences at treatment entry between opioid-dependent and cocaine-dependent males and females. Addictive Disorders and Their Treatment 3:110-121, 2004.
- [Background] Jones HE, Johnson RE, Bigelow GE, Silverman K, Mudric T, Strain EC. Safety and efficacy of L-tryptophan and behavioral incentives for treatment of cocaine dependence: a randomized clinical trial. Am J Addict. 2004 Oct-Dec;13(5):421-37. doi: 10.1080/10550490490512753. PMID 15764421